CLINICAL TRIAL: NCT07019662
Title: Comparing a Suture-based System for the Removal of Arterial and Veinous ECMO Cannulas to the Standard Approach
Acronym: CLOSE-ECMO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IHF GmbH - Institut für Herzinfarktforschung (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDR-004
Record Dates: First submitted 2025-05-26; First posted 2025-06-13 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: VA-ECMO

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decannulation using the Perclose™ ProStyle™ (Experimental)
  Interventions: Device: Decannulation with a medical device
- Standard of Care: Decannulation using surgical removal or manual compression (Active Comparator)
  Interventions: Procedure: Decannulation using surgical removal or manual compression

INTERVENTIONS:
Device: Decannulation with a medical device — Wound Closure with a medical device
  Arms: Decannulation using the Perclose™ ProStyle™
Procedure: Decannulation using surgical removal or manual compression — Wound closure using surgical removal or manual compression
  Arms: Standard of Care: Decannulation using surgical removal or manual compression

SUMMARY:
Background:

Patients with severe heart and lung failure may be treated with VA-ECMO (veno-arterial extracorporeal membrane oxygenation), a life-support machine that temporarily takes over the function of the heart and lungs. To connect the patient to ECMO, large tubes (cannulas) are inserted into major blood vessels in the groin area.

When the patient no longer needs ECMO, these cannulas must be removed - a process known as decannulation. Closing the artery after removing the cannula is a critical step and can be associated with complications such as bleeding, vessel injury, or blood clots.

Currently, there are different methods to close the artery:

* Surgical closure: open surgery to directly suture the artery
* Manual compression: pressing on the artery to stop bleeding
* Vascular closure devices (VCDs): special tools that close the artery through the skin

There is no clear standard yet on which method is safest and most effective for ECMO patients.

Purpose of the Study:

The study aims to determine whether using a vascular closure device is as safe and effective as the current standard methods for femoral artery closure after VA-ECMO.

Study Design:

This is a randomized controlled trial. Patients who are scheduled for decannulation after VA-ECMO support will be randomly assigned to one of two groups:

* Intervention Group: Patients receive a vascular closure device to seal the artery (Abbott Perclose™ ProStyle™ Suture-Mediated Closure System).
* Control Group: Patients receive standard care, which may be either:

  * Manual compression, or
  * Surgical closure, depending on the treating physician's judgment and the patient's condition.

This allows for a real-world comparison of the Closure Device method to current clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 Years
* Femoral placement of VA-ECMO with peripheral, percutaneous cannulation
* Arterial puncture site above the femoral bifurcation
* Cannula size must match or be smaller than the maximally licensed diameter for Perclose™ ProStyle™ (26 F (French) outer diameter arterial and 29 F outer diameter veinous)
* Patients must be eligible for either the Perclose™ ProStyle™ device or one of the two guideline-compliant alternatives for ECMO cannula removal (manual compression or surgical closure) according to the investigator's judgment.
* Initial arterial and/or venous puncture for ECMO cannulation was performed using ultrasound guidance with corresponding documentation available in the patient record.

Exclusion Criteria:

* Severe calcification
* Surgical cannulation
* Ongoing Infection of the ECMO site
* Any patient who does not fullfil the eligibility criteria for the use of the study device according to its current Instructions for Use (IFU), including known contraindications, limitations or warnings.
* Participation in another interventional clinical trial.
* Patients who are pregnant (assessed by clinical routine testing) or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of a combined vessel-orientated clinical endpoint (VOCE) | within 48 hours post ECMO removal

SECONDARY OUTCOMES:
Length of ICU (intensive care unit) stay post ECMO removal | Prior to hospital discharge, but no longer than 30 days after ECMO decannulation, whichever occurs first
Length of hospital stay post ECMO removal | Prior to hospital discharge, but no longer than 30 days after ECMO decannulation, whichever occurs first
Time to mobilization post ECMO removal | Prior to hospital discharge, but no longer than 30 days after ECMO decannulation, whichever occurs first
Costs of hospital stay | Prior to hospital discharge, but no longer than 30 days after ECMO decannulation, whichever occurs first
Incidence of Bleeding requiring transfusion (BARC3a) | At 48 hours post-ECMO and prior to hospital discharge, but no longer than 30 days after ECMO decannulation, whichever occurs first
Vascular complication requiring surgical or interventional therapy | At 48 hours post-ECMO and prior to hospital discharge, but no longer than 30 days after ECMO decannulation, whichever occurs first
Wound infection requiring antibiotic use or surgical debridement | At 48 hours post-ECMO and prior to hospital discharge, but no longer than 30 days after ECMO decannulation, whichever occurs first
Rate of pseudoaneurysms as detected by vascular Ultrasound | At 48 hours post-ECMO and prior to hospital discharge, but no longer than 30 days after ECMO decannulation, whichever occurs first
Rate of veinous thrombosis in the lower vessels as detected by vascular ultrasound | At 48 hours post-ECMO and prior to hospital discharge, but no longer than 30 days after ECMO decannulation, whichever occurs first
Rate of arterial thrombosis in the lower vessel as detected by vascular ultrasound | At 48 hours post-ECMO and prior to hospital discharge, but no longer than 30 days after ECMO decannulation, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Robert Stöhr, PD Dr. Dr., Principal Investigator — Universitäre Herz- und Gefäßzentrum Frankfurt ZIM - Med. Clinic 3 - Cardiology and Angiology
Locations (1):
- Universitäre Herz- und Gefäßzentrum Frankfurt ZIM - Med. Clinic 3 - Cardiology and Angiology, Frankfurt, Germany